CLINICAL TRIAL: NCT06228404
Title: The Safety and Efficacy Evaluation of Enhanced Autologous PSMA Chimeric Antigen Receptor T Cells in the Treatment of Refractory Castration Resistant Prostate Cancer
Brief Title: Clinical Study of Safety and Efficacy of Enhanced PSMA CAR- T in Refractory CRPC
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Bioray Laboratories (Industry)
Responsible Party: Principal Investigator, Ren Shancheng, Chief of Urology, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2022-BRL-501
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Castration-resistant Prostate Cancer; Castration-resistant Prostate Cancer
Keywords: Castration-resistant Prostate Cancer; Metastasis; Prostate-Speciﬁc Membrane Antigen; Chimeric Antigen Receptor T cell; Refractory Castration-resistant Prostate Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: A：0.25×106/kgBW B: 0.75×106/kgBW C: 2×106/kgBW
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enhanced autologous PSMA-CAR T: (Experimental): Enhanced autologous PSMA-CAR T is an electrotransfer system based on non-viral transposons that integrates the CAR gene into the genome of host cells by electrotransfer using PMSA as a target, while this CAR vector co-expresses enhanced factors and plays a strong regulatory role in innate and adaptive immunity.
  Interventions: Drug: Enhanced autologous PSMA-CAR T

INTERVENTIONS:
Drug: Enhanced autologous PSMA-CAR T — 3 escalated dosing cohorts are designed to explore safety and efficacy of enhanced autologous PSMA-CAR T:
  cohort A： CART-PSMA cells 0.25×106/kgBW, following lymphodepleting chemotherapy with cyclophosphamide 300 mg/m2/day and fludarabine 30 mg/m2/day given according to protocol;
  cohort B： CART-PSMA cells 0.75×106/kgBW，following lymphodepleting chemotherapy with cyclophosphamide 300 mg/m2/day and fludarabine 30 mg/m2/day given according to protocol;
  cohort C： CART-PSMA cells 2×106/kgBW，following lymphodepleting chemotherapy with cyclophosphamide 300 mg/m2/day and fludarabine 30 mg/m2/day given according to protocol;

SUMMARY:
This is one center, single-arm, open-label investigator initiated trial to assess the safety and efficacy of enhanced autologous PSMA chimeric antigen receptor T cells in the treatment for patients with refractory castration resistant prostate cancer, and the sample size is set to 7-18 subjects.

DETAILED DESCRIPTION:
This is one center, single-arm, open-label investigator initiated trial to assess the safety and efficacy of enhanced autologous PSMA chimeric antigen receptor T cells in the treatment for patients with refractory castration resistant prostate cancer, and the sample size is set to 7-18 subjects. Based on the "3 + 3" dose escalation design principle, subjects will be divided into 3 groups from low dose to high dose in sequence (Group A; Group B; Group C). Additional subjects will be enrolled into the RP2D group to ensure that 6-9 efficacy-evaluable subjects are available in the RP2D group before entering the phase II study.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understood and voluntarily signed informed consent for this study;
2. male, aged 18-75 years;
3. expected survival of more than 6 months;
4. metastatic castration-resistant prostate adenocarcinoma (CRPC) patients.
5. Receiving CRPC standard treatment (such as new endocrine therapy, chemotherapy and radium-223, etc., one or more of the combination therapy) after the diagnosis of CRPC, ineffective or progressive disease (PSA continued to rise for 3 months, or bone scan/whole-body MRI/PET-CT showed local recurrence or new metastatic lesions, demonstrating disease progression);
6. PSMA expression in tumor cells was positive in immunohistochemical staining of prostate/metastatic biopsy tissue before enrollment;
7. ECOG score < 2 ;
8. virological examination HAV (hepatitis A virus), HBV (hepatitis B virus), HCV (hepatitis C virus), HIV (human immunodeficiency virus), TP (Treponema pallidum) quantitative detection was negative, (antigen and antibody screening method unknown, confirmed by nucleic acid method); hematological parameters met the following criteria: a. hemoglobin > 100 g/L; b. platelet count > 100 × 109/L; c. neutrophils > 1.5 × 109/L.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria will be excluded:

1. have received any previous treatment with CAR-T therapy ;
2. have received any previous treatment that targets PSMA;
3. tumor pathology suggests a special type of prostate cancer (e.g., neuroendocrine prostate cancer, etc.)
4. severe mental disorders;
5. suffered from previous malignancies, except for the following: a. basal cell carcinoma or squamous cell carcinoma after standardized treatment; b. having a primary malignancy, but completely resected, with a complete remission time of ≥ 5 years.
6. Subjects with severe cardiovascular disease; a.New York Heart Association (NYHA) stage III or IV congestive heart failure; b.Myocardial infarction ≤ 6 months prior to enrollment or coronary artery bypass graft (CABG); c.Clinically significant ventricular arrhythmia, or history of unexplained syncope, nonvasovagal or not due to dehydration; d.History of severe non-ischemic cardiomyopathy; e.Decreased left ventricular ejection fraction (LVEF < 55%) as assessed by echocardiogram or multigated acquisition (MUGA) scan, abnormal interventricular septal thickness and atrioventricular size associated with myocardial amyloidosis;
7. active infectious disease or any major infectious event requiring high grade antibiotics;
8. organ function in the following abnormalities: a. serum aspartate aminotransferase or alanine aminotransferase > 2.5ULN; CK > ULN; CK-MB > ULN; TnT > 1.5ULN; b. total bilirubin > 1.5ULN; c. partial prothrombin time or activated partial thromboplastin time or international normalized ratio > 1.5ULN in the absence of anticoagulant therapy;
9. participation in other clinical studies in the past three months or previous treatment with any gene therapy product;
10. intolerance or hypersensitivity to cyclophosphamide and fludarabine chemotherapy;
11. unsuitability to participate in this clinical study in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-03-03 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
DLT | Within 28 Days After Enhanced autologous PSMA-CAR T Infusion
  The number and severity of dose-limiting toxicity (DLT) events

SECONDARY OUTCOMES:
PSA response rate | From 3 weeks to 6 months after Enhanced autologous PSMA-CAR T infusion
  PSA50 response, PSA90 response: PSA response determined as ≥ 50% or ≥ 90% reduction in PSA level from baseline to post-baseline and reassessed at least 3 weeks later
ORR | 6 months after Enhanced autologous PSMA-CAR T infusion
  Objective response rate ORR = CR + PR

CONTACTS AND LOCATIONS:
Locations (1):
- Changzheng hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No